CLINICAL TRIAL: NCT05013216
Title: Mutant KRAS -Targeted Long Peptide Vaccine for Patients at High Risk of Developing Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Stand Up To Cancer (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: J2177; IRB00288752 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: High Risk Cancer; Pancreatic Cancer
Keywords: KRAS Peptide Vaccine; Neoantigen Vaccines; Cancer Vaccines; Immunotherapy; Pancreatic Ductal Adenocarcinoma (PDAC)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Patients at high risk of developing pancreatic cancer. (Experimental): Patients will include those who have undergone pancreatic imaging with MRI or CT or EUS and found to have one or more pancreatic imaging abnormalities such as a pancreatic cyst consistent with an intraductal papillary mucinous neoplasm (IPMN) or parenchymal changes consistent with pancreatic intraepithelial neoplasia (PanIN). additionally patients with:
  1. familial pancreatic cancer relatives
  2. germline mutation carriers with an estimated lifetime risk of pancreatic cancer of ~10% or higher
  3. germline mutation carriers with an estimated lifetime risk of pancreatic cancer of ~5%, all detailed in Section 3.1.1. These patients must also (as defined in Section 3.1.2).
  Interventions: Drug: Cohort A: Patients at high risk of developing pancreatic cancer.
- Cohort B: Patients must have evidence of a pancreatic cystic neoplasm (Experimental): Patients must have clinical, radiographic, or histologic evidence of a pancreatic cystic neoplasm with high-risk features warranting surgical resection per the discretion of the treating hepatobiliary surgeon. In addition, cyst fluid analysis must demonstrate the presence of one of the six KRAS mutations included in the study vaccine. Germline mutation testing or a positive family history of pancreatic cancer is not required for enrollment in Cohort B.
  Interventions: Drug: Cohort B: Patients must have evidence of a pancreatic cystic neoplasm

INTERVENTIONS:
Drug: Cohort A: Patients at high risk of developing pancreatic cancer. — 1. KRAS peptide vaccine with poly-ICLC adjuvant will be administered on Prime week 1, 3, and 5. Boost vaccinations with will be administered at week 13. All subjects will return to the study site approximately 28 days (+ 7 days) after the last vaccination for an End of Treatment (EOT) and safety evaluation.
  2. Drug: up to 1.8 mg KRAS peptide vaccine + 0.5mg Poly-ICLC
  Other Names: Hiltonol® (Poly-ICLC)
  Arms: Cohort A: Patients at high risk of developing pancreatic cancer.
Drug: Cohort B: Patients must have evidence of a pancreatic cystic neoplasm — Patients will receive KRAS peptide vaccine with poly-ICLC adjuvant as two prime vaccinations on weeks 1 and 2. Surgery is considered standard of care. Surgery will occur at the discretion of the treating hepatobiliary surgeon and is not dictated by this protocol. Subjects will return to the study site approximately at week 4 (+ 7 days) for a safety evaluation prior to surgery. Subjects will have an End of Treatment (EOT) visit at study Week 8 (+ 7 days).
  Other Names: Hiltonol® (Poly-ICLC)
  Arms: Cohort B: Patients must have evidence of a pancreatic cystic neoplasm

SUMMARY:
This Phase 1 study will evaluate safety and the immune response to pooled mutant-KRAS peptide vaccine with poly-ICLC adjuvant for patients who have been identified to be at risk of developing pancreatic cancer.

DETAILED DESCRIPTION:
This study will evaluate safety and the immune response to pooled mutant-KRAS peptide vaccine (KRAS peptide vaccine) with poly-ICLC adjuvant. The primary endpoints of this study are to determine the safety of administering the KRAS peptide vaccine with poly-ICLC adjuvant and to assess the maximal percent change of IFN-γ-producing mutant-KRAS-specific T cells per patient at any time after vaccination. Twenty five patients will be enrolled to achieve 20 evaluable patients for Cohort A. Twelve patients will be enrolled to achieve 10 evaluable patients for Cohort B.

For all patients, the study will consist of a screening phase, treatment phase, and a follow-up visit. All subjects will have the option remaining on study with annual follow-up visits that begin approximately one year after the last vaccine dose and continue annually thereafter until study closure.

ELIGIBILITY:
Inclusion Criteria:

Cohort A: Must fall into one of the three categories defined as high risk of developing pancreatic cancer and are undergoing pancreatic surveillance AND 2) have documented radiographic evidence of a pancreatic abnormality such as a pancreatic cyst.

* High Risk Group 1 (familial pancreatic cancer relatives):

  * >/=55 years old or 10 years younger than the age of youngest relative with pancreatic cancer, and
  * Come from a family with 2 or more members with a history of pancreatic cancer (2 of which have a first-degree relationship consistent with familial pancreatic cancer), and
  * Have a first-degree relationship with at least one of the relatives with pancreatic cancer.
  * If there are 2 or more affected blood relatives, at least 1 must be a first-degree relative of the individual being screened.
* High Risk Group 2 (Germline mutation carriers with an associated with an estimated lifetime risk of pancreatic cancer of ~10% or higher):

  * >/=40 years old and the Patient is a carrier of FAMMM (p16/CDKN2A) mutation regardless of family pancreas cancer history.

OR

* >/= 50 years old or 10 years younger than the age of the youngest relative with pancreatic cancer, and the Patient is a carrier of a known BRCA2, ATM, PALB2 mutation.
* Persons with known genetic mutation should have proof of mutation status. Those who had research-related genetic testing must have confirmation by a clinical CLIA-certified laboratory.

  o High Risk Group 3 (Germline mutation carriers with an associated with an estimated lifetime risk of pancreatic cancer of ~5%):
* >/= 50 years old or 10 years younger than the age of the youngest relative with pancreatic cancer, and
* The patient is a carrier of a known, BRCA1, or HNPCC (hereditary non-polyposis colorectal cancer or Lynch syndrome, hMLH1, hMSH2, PMS1, hMSH6, EpCAM) gene mutation, and there is > 1 pancreatic cancer in the family, one of whom is a first- or second-degree relative of the subject to be screened.
* Persons with known genetic mutation should have proof of mutation status. Those who had research-related genetic testing must have confirmation by a clinical CLIA-certified laboratory.
* Cohort A: Patients must have a pancreatic imaging abnormality that is being followed by pancreatic imaging surveillance (EUS and/or MRI and /or CT), such as a pancreatic cyst consistent with an IPMN or parenchymal abnormalities consistent with PanIN.

  * Cohort B: Patients must have clinical, radiographic, or histologic evidence of pancreatic cystic neoplasm with high-risk features warranting surgical resection per the discretion of the treating hepatobiliary surgeon.
  * Cohort B: Patients must have cystic fluid testing that demonstrates the presence of one of the six KRAS mutations included in the study vaccine.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Ability to understand and willingness to sign a written informed consent document.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.

Exclusion Criteria:

* If expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Within 4 weeks prior to first dose of study drug.

  o Any systemic or topical corticosteroids at immunosuppressive agents.
* Within 4 weeks prior to first dose of study drug.

  * Any investigational device.
  * Has received a live vaccine.
  * Received any allergen hyposensitization therapy.
  * Any major surgery.
* Infection with HIV or hepatitis B or C.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements monoclonal antibody.
* Has a diagnosis of immunodeficiency.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Unwilling or unable to follow the study schedule for any reason.
* Are pregnant or breastfeeding.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing study drug-related toxicities | 1.5 years
  Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0
Maximal percentage of change of interferon (IFN-γ) producing mutant-KRAS-specific CD8 and CD4 T cells | 17 weeks
  Maximal percent change per patient within 17 weeks after vaccination.

SECONDARY OUTCOMES:
Fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 5 weeks. | Baseline, 5 weeks (Cohort A)
  Evaluated by the fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 5 weeks after vaccination compared to pre-vaccination baseline.
Fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 13 weeks. | Baseline, 13 weeks (Cohort A)
  Evaluated by the fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 13 weeks after vaccination compared to pre-vaccination baseline.
Fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 17 weeks. | Baseline,17 weeks (Cohort A)
  Evaluated by the fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 17 (EOT) weeks after vaccination compared to pre-vaccination baseline.

OTHER OUTCOMES:
Fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 1 weeks. | Baseline, 1 week (Cohort B)
  Evaluated by the fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 5 weeks after vaccination compared to pre-vaccination baseline.
Fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 4 weeks. | Baseline, 4 weeks (Cohort B)
  Evaluated by the fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 13 weeks after vaccination compared to pre-vaccination baseline.
Fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 8 weeks. | Baseline, 8 weeks (Cohort B)
  Evaluated by the fold change in interferon-producing mutant-KRAS-specific CD8 and CD4 T cells at 17 (EOT) weeks after vaccination compared to pre-vaccination baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at the Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No